CLINICAL TRIAL: NCT02063945
Title: The Assessment of Efficacy and Tolerability of Methylphenidate vs. Risperidone in the Treatment of Children and Adolescents With ADHD and Disruptive Disorders
Brief Title: Methylphenidate vs. Risperidone for the Treatment of Children and Adolescents With ADHD and Disruptive Disorders
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Major difficulties recruiting participants
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Doron Gothelf MD, Head of child and adolescent psychiatry unit, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-13-0564-DG-CTIL
Record Dates: First submitted 2014-02-11; First posted 2014-02-17 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Attention Deficit/Hyperactivity Disorder; Oppositional Defiant Disorder; Conduct Disorder
Keywords: ADHA; ODD; Conduct disorder; Aggression; Treatment; Methylphenidate; Risperidone
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder; Conduct Disorder; Aggression | interventions — Methylphenidate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylphenidate (Active Comparator): Participants in this arm will be given either "Concerta" - a long acting (12 hours) Methylphenidate pill - once daily, in the morning (starting dose 1 mg/kg, max dose 2 mg/kg), or "Ritalin LA" - a long acting (10 hours) Methylphenidate pill - once daily, in the morning (starting dose 0.6 mg/kg, max dose 1.5 mg/kg) for children who can not swallow pills.
  Interventions: Drug: Methylphenidate
- Risperidone (Active Comparator): Participants in this arm will be given a low dose of Risperidone. Starting dose will be 0.5 mg/d, max dose will be 2 mg/d.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Methylphenidate — As stated in arm/group
  Other Names: Ritalin; Ritalin SR; Ritalin LA; Concerta
  Arms: Methylphenidate
Drug: Risperidone — As stated in arm/group
  Other Names: Risperdal
  Arms: Risperidone

SUMMARY:
Attention Deficit/Hyperactivity Disorder (ADHD) is one the most prevalent mental disorders among children and adolescents, with a prevalence of 5% in western culture. The basics of the disorder: inattentive and hyperactive/impulsive behaviors that manifest in a variety of settings causing a dysfunction in everyday life. ADHD can be subdivided into three sub-types: predominantly inattentive, predominantly hyperactive/impulsive or combined type. Common co-morbidities of ADHD are disruptive disorders; Oppositional defiant disorder (ODD) being the major one with about half of children with the combined sub-type ADHD and about a quarter of children with the predominantly inattentive also suffering from ODD. Conduct disorder is a co-morbidity for about a quarter of children with the combined sub-type ADHD. The co-occurrence of these disorders is thought to have a negative effect on the outcome of both of them.

Methylphenidate (MPH), short or long acting, is the mainstay of medical treatment for ADHD patients, it's efficacy proven in a variety of studies. It should be noted that MPH has also been proven to have a beneficial effect on children with disruptive behaviors. For children with disruptive disorders Risperidone is the mainstay of medical treatment, and has been proven in clinical trials.

To the best of their knowledge, a "head to head" study comparing these two drugs for the treatment of pediatric patients with ADHD and co-morbidity of disruptive disorders was never done before. The investigators aim is to examine the efficacy and tolerability of MPH vs. Risperidone in this population. In addition, the investigators will apply DSM5's cross cutting symptom measures scales is order to further define this unique subset of patients.

Disruptive mood dysregulation disorder (DMDD) is a new diagnosis in the latest version of the diagnostic and statistical manual (DSM5). It's main features: sever recurrent temper outbursts that are inconsistent with developmental level and occur on average three times a week, the outbursts occur in at least two settings and the mood between outbursts is irritable or angry. This diagnosis is in the differential diagnosis of ADHD with disruptive disorders.

DETAILED DESCRIPTION:
Secondary study aims:

1. Comparing the efficacy and tolerability of MPH vs. Risperidone in the treatment of depressive symptoms in children and adolescents with ADHD and disruptive disorders.
2. Comparing the efficacy and tolerability of MPH vs. Risperidone in the treatment of manic symptoms in children and adolescents with ADHD and disruptive disorders.
3. Comparing the impact of MPH vs. Risperidone on overall every day functioning of children and adolescents with ADHD and disruptive disorder.
4. Comparing the impact of MPH vs. Risperidone on nighttime sleep of children and adolescents with ADHD and disruptive disorder.
5. Comparing the impact of MPH vs. Risperidone on weight and height of children and adolescents with ADHD and disruptive disorder.
6. Assessing the overlap between the diagnosis of ADHD and disruptive disorders and DMDD.
7. Assessing mood disorders and response to MPH vs. Risperidone treatment in children and adolescents with ADHD and disruptive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ADHD (any sub-type) with oppositional defiant disorder.
* Clinical diagnosis of ADHD (any sub-type) with conduct disorder.
* Clinical diagnosis of other specified ADHD with oppositional defiant disorder.
* Clinical diagnosis of other specified ADHD with conduct disorder.
* Clinical diagnosis of unspecified ADHD with oppositional defiant disorder.
* Clinical diagnosis of unspecified ADHD with conduct disorder.

Exclusion Criteria:

* Participant who do not qualify for inclusion criteria.
* Participant who are not willing to join the study.
* Epilepsy.
* Neuro-genetic syndromes.
* Brain tumors.
* Autism.
* Participants who are under psychiatric medication and have changed it (dose or kind) in the last month.
* Congenital heart, kidney of liver defects.
* Cardiomyopathies.
* Past hypersensitivity to Methylphenidate or Risperidone.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of aggressive behaviors. | baseline, 2 weeks, 4 weeks, 8 weeks.
  The Retrospective Modified Overt Aggression Scale (R-MOAS) will be used for the the assessment of aggressive behaviors and their response to treatment.

SECONDARY OUTCOMES:
Clinical Global Impression - Improvement scale (CGI-I) questionnaire | 2 weeks, 4 weeks, 8 weeks.
  The Clinical Global Impression - Improvement scale (CGI-I) is a scale used for the assessment of overall symptom change.
ADHD-RS questionnaire | baseline, 2 weeks, 4 weeks, 8 weeks.
  The ADHD Rating Scale (ADHD-RS) is a routinely use questionnaire used for the assessment of ADHD symptomatology and it's response to treatment.
Children's Depression Rating Scale (CDRS) questionnaire | baseline, 2 weeks, 4 weeks, 8 weeks.
  The Children's Depression Rating Scale (CDRS) is a routinely use questionnaire used for the assessment of depression symptomatology and it's response to treatment.
Young Mania Rating Scale (YMRS) questionnaire | baseline, 2 weeks, 4 weeks, 8 weeks.
  The Young Mania Rating Scale (YMRS) is a routinely use questionnaire used for the assessment of mania symptomatology and it's response to treatment.
Children Sleep Habits Questionnaire (CSHQ) | baseline, 2 weeks, 4 weeks, 8 weeks.
  The Children Sleep Habits Questionnaire (CSHQ) is a routinely use questionnaire used for the assessment of children sleep habits.
Clinical Global Impression - Severity (CGI-S) questionnaire | baseline, 2 weeks, 4 weeks, 8 weeks.
  The Clinical Global Impression - Severity scale (CGI-S) is a scale used for the assessment of overall symptom severity.

OTHER OUTCOMES:
Height and Weight | baseline, 2 weeks, 4 weeks, 8 weeks.
Blood Tests | baseline, 8 weeks.
  Electrolytes, liver function tests, creatinine, Prolactin, complete blood count.

CONTACTS AND LOCATIONS:
Overall Officials: Doron Gothelf, professor, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Connor DF, Steeber J, McBurnett K. A review of attention-deficit/hyperactivity disorder complicated by symptoms of oppositional defiant disorder or conduct disorder. J Dev Behav Pediatr. 2010 Jun;31(5):427-40. doi: 10.1097/DBP.0b013e3181e121bd. PMID 20535081
- [Background] Hodgkins P, Shaw M, Coghill D, Hechtman L. Amfetamine and methylphenidate medications for attention-deficit/hyperactivity disorder: complementary treatment options. Eur Child Adolesc Psychiatry. 2012 Sep;21(9):477-92. doi: 10.1007/s00787-012-0286-5. Epub 2012 Jul 5. PMID 22763750
- [Background] Subcommittee on Attention-Deficit/Hyperactivity Disorder; Steering Committee on Quality Improvement and Management; Wolraich M, Brown L, Brown RT, DuPaul G, Earls M, Feldman HM, Ganiats TG, Kaplanek B, Meyer B, Perrin J, Pierce K, Reiff M, Stein MT, Visser S. ADHD: clinical practice guideline for the diagnosis, evaluation, and treatment of attention-deficit/hyperactivity disorder in children and adolescents. Pediatrics. 2011 Nov;128(5):1007-22. doi: 10.1542/peds.2011-2654. Epub 2011 Oct 16. PMID 22003063
- [Background] Seida JC, Schouten JR, Boylan K, Newton AS, Mousavi SS, Beaith A, Vandermeer B, Dryden DM, Carrey N. Antipsychotics for children and young adults: a comparative effectiveness review. Pediatrics. 2012 Mar;129(3):e771-84. doi: 10.1542/peds.2011-2158. Epub 2012 Feb 20. PMID 22351885
- [Background] Poznanski EO, Cook SC, Carroll BJ. A depression rating scale for children. Pediatrics. 1979 Oct;64(4):442-50. PMID 492809
- [Background] Youngstrom EA, Danielson CK, Findling RL, Gracious BL, Calabrese JR. Factor structure of the Young Mania Rating Scale for use with youths ages 5 to 17 years. J Clin Child Adolesc Psychol. 2002 Dec;31(4):567-72. doi: 10.1207/S15374424JCCP3104_15. PMID 12402575
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Background] Harris S, Oakly C, Picchioni M. Quantifying Violence in Mental Health Research. Aggression and Violent Behavior 18(6):695-701, 2013.
- [Background] Armenteros JL, Lewis JE, Davalos M. Risperidone augmentation for treatment-resistant aggression in attention-deficit/hyperactivity disorder: a placebo-controlled pilot study. J Am Acad Child Adolesc Psychiatry. 2007 May;46(5):558-565. doi: 10.1097/chi.0b013e3180323354. PMID 17450046